CLINICAL TRIAL: NCT04186117
Title: Clinical and Biological Evaluation to Caracterize Circulating Tumoral Cells in Colorectal Cancer
Brief Title: Development of Clinical and Biological Database in Colorectal Cancer
Acronym: CIRCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: URC 2015/16
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colon Cancer
Keywords: colon cancer; circulating tumoral cells
MeSH Terms: conditions — Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all the patients include in the study :
  - Blood samples collected at before any treatment
  In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample before any treatment

SUMMARY:
Creation of circulating cancer cell-lines and caracterisation of these cell-lines which will be collected before any treatment in patients with metastatic colon adenocarcinoma

DETAILED DESCRIPTION:
In the light of literature data, it becomes crucial to develop models for studying the functionality of CTCs. In this context, xenograft models in nude mice have recently been described9,10. Establishing cell lines to allow CTC amplification to have enough material to work is an attractive approach. Some recent studies have demonstrated the feasibility of establishing such tools in breast or prostate cancer, 11, 12 but no studies have been done for colorectal cancer. Thus on the basis of the hypothesis that circulating tumor cells could be, or at least contain, cancerous stem cells, we propose to isolate them under conditions that promote their survival in order to characterize them in the particular context of colorectal cancer.

If CTCs consist at least in part of CSCs, they should survive in an environment favorable to the culture of these cells. It is for this reason that purified CTCs will be seeded in plaques that prevent cell adhesion and in a serum-free medium but including growth factors (M12) under hypoxia conditions to approximate their original context. The ability of these cells to form spheres will be observed under these conditions.

In this context, the team of the Institute of Functional Genomics of Montpellier are the first, to have developed and characterized three lines of CTC from blood samples of patients with metastatic colon cancer (Grillet F. and al; submitted for publication). In addition to the characterization of these rare cells and the decryption of some of the mechanisms involved in tumor dissemination, this tool is very valuable for the clinic. Indeed, it could help the establishment of personalized medicine to test quickly (less than 3 weeks) on the CTC of the patient, the effectiveness of conventional treatments but also new drugs included in clinical protocols. For the basic research part, this line will help us to characterize these cells because the number is no longer a limiting factor, the main objective now being to obtain more lines from a blood sample from patients with different profiles by optimizing cell culture conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years
* Histological evidence of metastatic colorectal cancer
* Naïve patients receiving chemotherapy at the metastatic stage or who have received adjuvant chemotherapy for more than 6 months
* Obtain signed informed consent prior to any specific preselection procedure.

Exclusion Criteria:

* History of Chemotherapy Treatment and / or Targeted Therapy for Metastatic Colorectal Cancer
* Breastfeeding or pregnant woman
* Patient whose regular follow-up is impossible for psychological, family, social or geographical reasons
* Any severe or unstable medical, psychiatric or other condition that may interfere with the patient's safety, consent or compliance with the study protocol
* Patient not benefiting from a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Isolation of circulating tumoral cells | Until the study completion : 54 months
  among 100 patients, to isolate at least 10 cell-lines to show the heterogeneity between patients

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- ICM Val d'Aurelle, Montpellier, France